CLINICAL TRIAL: NCT07191405
Title: The Efficacy and Safety of Chemotherapy and Immune Therapy Combined With Lactobacillus Johnsonii in Patients With Metastatic or Locally Advanced Unresectable or Recurrent EGFR/ALK Wild-type Adenocarcinoma Non-small Cell Lung Cancer (NSCLC), PD-L1 Positive (CPS≥1) Triple-negative Breast Cancer (TNBC) and HER2-negative Gastric or Gastro-oesophageal Junction Adenocarcinoma: a Multicenter, Randomized, Double-blind, Clinical Trial.
Brief Title: Clinical Study of Chemotherapy and Immunotherapy Combined With Lactobacillus Johnsonii in Patients With Multiple Irresectable Solid Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1242
Record Dates: First submitted 2025-07-10; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-06

CONDITIONS: Immunotherapy; Chemotherapy
Keywords: Lactobacillus johnsonii; Immunotherapy; Chemotherapy; unresectable or recurrent EGFR/ALK wild-type NSCLC; PD-L1 positive TNBC; HER2-negative gastric or gastro-oesophageal junction adenocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Subgroup A: Experimental arm (Experimental): This arm will include 24 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent EGFR/ALK wild-type adenocarcinoma non-small cell lung cancer (NSCLC). The treatment regimen consists of chemotherapy combined with immunotherapy tislelizumab (200 mg IV on Day 1) + pemetrexed (500 mg/m² BSA IV on Day 1) + cisplatin (75 mg/m² BSA IV on Day 1)+oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily). Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily)
- Subgroup A: Control arm (Placebo Comparator): This arm will include 24 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent EGFR/ALK wild-type adenocarcinoma non-small cell lung cancer (NSCLC). The treatment regimen consists of chemotherapy combined with immunotherapy tislelizumab (200 mg IV on Day 1) + pemetrexed (500 mg/m² BSA IV on Day 1) + cisplatin (75 mg/m² BSA IV on Day 1)+ placebo orally twice daily. Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: Placebo
- Subgroup B: Experimental arm (Experimental): This arm will include 26 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent PD-L1-positive (CPS ≥1) triple-negative breast cancer (TNBC). The treatment regimen consists of toripalimab (240 mg IV on Day 1) + nab-paclitaxel (260 mg/m² BSA IV on Day 1) + carboplatin (300 mg/m² BSA IV on Day 1) + oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily). Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily)
- Subgroup B: Control arm (Placebo Comparator): This arm will include 26 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent PD-L1-positive (CPS ≥1) triple-negative breast cancer (TNBC). The treatment regimen consists of toripalimab (240 mg IV on Day 1) + nab-paclitaxel (260 mg/m² BSA IV on Day 1) + carboplatin (300 mg/m² BSA IV on Day 1) + placebo orally twice daily. Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: Placebo
- Subgroup C: Experimental arm (Experimental): This arm will include 28 patients with metastatic or locally advanced unresectable or recurrent HER2-negative gastric or gastroesophageal junction adenocarcinoma. The treatment regimen consists of tislelizumab (200 mg IV on Day 1) + oxaliplatin (130 mg/m² BSA IV on Day 1) + capecitabine (1000 mg/m² BSA orally twice daily, taken 30 minutes after meals on Days 1-14) + oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily). Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily)
- Subgroup C: Control arm (Placebo Comparator): This arm will include 28 patients with metastatic or locally advanced unresectable or recurrent HER2-negative gastric or gastroesophageal junction adenocarcinoma. The treatment regimen consists of tislelizumab (200 mg IV on Day 1) + oxaliplatin (130 mg/m² BSA IV on Day 1) + capecitabine (1000 mg/m² BSA orally twice daily, taken 30 minutes after meals on Days 1-14) + placebo orally twice daily. Tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily) — Lactobacillus johnsonii, as a member of gut probiotics, has recently gained attention for its potential role in tumor immunotherapy due to its ability to modulate the immune system and maintain gut microbiota balance. Below is a summary of its possible mechanisms and applications: 1.Modulating Gut Microbiota and Immune Microenvironment. 2.Direct or Indirect Activation of Anti-Tumor Immunity. 3.Enhancing Efficacy of Immune Checkpoint Inhibitors (ICIs) . 4.Anti-Tumor Effects of Microbial Metabolites. 5.Preclinical and Clinical Research Progress.
  Arms: Subgroup A: Experimental arm; Subgroup B: Experimental arm; Subgroup C: Experimental arm
Dietary Supplement: Placebo — oral take placebo twice a day
  Arms: Subgroup A: Control arm; Subgroup B: Control arm; Subgroup C: Control arm

SUMMARY:
This study plans to enroll 156 patients aged 18-75, who will be randomly divided into two groups to evaluate the clinical efficacy and safety of chemotherapy and immune therapy combined with Lactobacillus johnsonii in patients with various advanced unresectable tumors.

This study was divided into three subgroups, with 48,52 and 56 subjects in each group respectively，randomly assigned to the experimental or control group in a 1:1 ratio.

Subgroup A will include 48 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent EGFR/ALK wild-type adenocarcinoma non-small cell lung cancer (NSCLC). The treatment regimen consists of chemotherapy combined with immunotherapy tislelizumab (200 mg IV on Day 1) + pemetrexed (500 mg/m² BSA IV on Day 1) + cisplatin (75 mg/m² BSA IV on Day 1). The experimental group will additionally receive oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily), while the control group will receive a placebo orally twice daily. Standard tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.

Subgroup B will include 52 patients with histologically or cytologically confirmed metastatic or locally advanced unresectable or recurrent PD-L1-positive (CPS ≥1) triple-negative breast cancer (TNBC). The treatment regimen consists of toripalimab (240 mg IV on Day 1) + nab-paclitaxel (260 mg/m² BSA IV on Day 1) + carboplatin (300 mg/m² BSA IV on Day 1). The experimental group will additionally receive oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily), while the control group will receive a placebo orally twice daily. Standard tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.

Subgroup C will include 56 patients with metastatic or locally advanced unresectable or recurrent HER2-negative gastric or gastroesophageal junction adenocarcinoma. The treatment regimen consists of tislelizumab (200 mg IV on Day 1) + oxaliplatin (130 mg/m² BSA IV on Day 1) + capecitabine (1000 mg/m² BSA orally twice daily, taken 30 minutes after meals on Days 1-14). The experimental group will additionally receive oral Lactobacillus johnsonii (1×10¹¹ CFU, twice daily), while the control group will receive a placebo orally twice daily. Standard tumor treatment will be administered every 3 weeks, with follow-up every 6 weeks to assess treatment efficacy and drug-related adverse reactions. Follow-up time points: 0, 6, 12, 18, and 24 weeks.

Primary Efficacy Endpoint: Progression-Free Survival (PFS): Time from randomization to tumor progression or death from any cause (whichever occurs first).

Secondary Efficacy Endpoints:

1. Changes in gut microbiome composition in stool samples: qPCR and 16sRNA analysis of microbial composition, including Lactobacillus johnsonii, immunotherapy-related bacterial abundance, and microbial diversity.
2. Changes in immune cell subsets in blood, just like Tregs, MDSCs, CD8+ T cells.
3. Changes in blood levels of IL-6, IL-8, and other cytokines/chemokines.
4. Changes in blood indole derivatives, for example, indolepropionic acid.
5. Characterization of the tumor microenvironment in archived tumor samples.
6. Objective Response Rate (ORR): Proportion of patients with tumor shrinkage meeting predefined criteria and sustained for a minimum duration (CR + PR).
7. Disease Control Rate (DCR): Percentage of evaluable cases achieving response (PR+CR) or stable disease (SD).
8. Duration of Response (DOR): Time from first objective response to disease progression (PD) or death before PD, reflecting the durability of ORR.
9. Disease Control Rate (DCR): Percentage of evaluable cases achieving response (PR+CR) or stable disease (SD).
10. Overall Survival (OS): Time from randomization to death from any cause.
11. Percentage of patients with immune checkpoint inhibitor-related adverse events (irAEs).

DETAILED DESCRIPTION:
Research Objective This study is a randomized, double-blind, controlled, prospective multicenter clinical trial, designed to evaluate the clinical efficacy and safety of chemotherapy and immune therapy combined with Lactobacillus johnsonii in patients with various advanced unresectable solid tumors.

Study Methods:

Design: Randomized, controlled, double-blind, multicenter clinical study. Duration: 6-12 months. Start Date: Upon ethical approval and completion of clinical trial registration.

Study Design:

1. Overall Design:

   A prospective, multicenter, randomized controlled trial assessing the efficacy and safety of immunotherapy supplemented with Lactobacillus johnsonii in various tumor types.

   Eligible patients will be randomly assigned to treatment groups after screening.

   Participating Centers:

   The Second Affiliated Hospital, Zhejiang University School of Medicine Zhejiang Cancer Hospital Hangzhou First People's Hospital The First Affiliated Hospital of Wenzhou Medical University
2. Sample Size Calculation:

   Statistical Parameters: Two-sided test, α=0.05, power (1-β)=80%.

   Sample Size per subgroup:

   Subgroup A (Lung cancer): 48 cases (24 per group) Subgroup B (Breast cancer): 52 cases (26 per group) Subgroup C (Gastric/gastroesophageal junction adenocarcinoma): 56 cases (28 per group) Total Sample Size: 156 cases (calculated using PASS 15 software).
3. Randomization:

   Computer-generated random sequences (1:1 allocation). Managed by independent researchers to avoid bias. Each participant receives a unique screening number (non-reusable, even if withdrawn).
4. Study Population:

Inclusion Criteria:

1. Signed informed consent.
2. Age 18-75 years.
3. Histologically confirmed unresectable/metastatic tumors:

   EGFR/ALK wild-type adenocarcinoma non-small cell lung cancer (NSCLC) PD-L1+ (CPS≥1) triple-negative breast cancer (TNBC) HER2- gastric/gastroesophageal adenocarcinoma
4. ≥1 measurable lesion (RECIST v1.1).
5. Progression after PD-1/PD-L1 inhibitor therapy (defined as:

   - ≥2 doses administered.
   * Radiographic progression per RECIST/iRECIST/irRECIST, confirmed ≥4 weeks later.
   * Progression within 12 weeks of last PD-1/PD-L1 dose.
6. Adequate organ function.
7. ECOG performance status 0-1.
8. Negative pregnancy test (urine/serum β-HCG) for women of childbearing potential.

Exclusion Criteria

Subjects meeting any of the following will be excluded:

1. Prior allogeneic transplantation (cells, tissues, or solid organs).
2. History of immune-related adverse events (irAEs) from immunomodulators (e.g., PD-1/PD-L1 or CTLA-4 inhibitors) leading to permanent discontinuation or Grade 3/4 severity.
3. Recent anticancer therapy (chemotherapy/immunotherapy/biologics/experimental drugs) within: <5 half-lives of the drug or <21 days before starting study treatment (whichever is shorter). Exceptions: Stable hormone therapy (e.g., for prostate/breast/ovarian cancer).
4. Concomitant corticosteroid use (>10 mg prednisone/day or equivalent) within 7 days prior to treatment, unless for physiological replacement (≤10 mg/day) or non-immunosuppressive purposes (e.g., inhaled/topical steroids).
5. Severe cardiac dysfunction, including: NYHA Class III-IV heart failure, symptomatic coronary artery disease, severe ventricular arrhythmias, myocardial infarction/unstable angina within 6 months.
6. Active autoimmune disease requiring systemic treatment (immunosuppressants/corticosteroids) in the past 2 years, except: Hormone replacement (thyroxine, insulin, physiologic corticosteroids).
7. Active severe infection requiring systemic therapy.
8. Antibiotic use completed within 2 weeks before the first dose.
9. Psychiatric or substance abuse disorders compromising protocol compliance.
10. Live vaccines administered within 28 days before treatment.
11. Active HIV or hepatitis (A/B/C) infection.
12. History of steroid-requiring (non-infectious) pneumonitis or current active pneumonitis.
13. Other malignancies requiring active treatment or progressing within 2 years (exceptions: Non-melanoma skin cancer, cervical/prostate carcinoma in situ).
14. Pregnancy or lactation.
15. Known intolerance/allergy to study drugs.
16. Other conditions deemed unsuitable by investigators.

3. Subject Discontinuation/Withdrawal

- Pre-randomization withdrawal: Considered a screen failure; reasons must be documented in medical records.

* Post-enrollment withdrawal:
* Subjects may withdraw at any time without penalty or loss of benefits.
* Reasons (if provided) should be recorded (e.g., intolerable AEs, consent withdrawal).
* Protocol-defined discontinuation if:

  1. Use of prohibited immunomodulatory drugs. 2. Pregnancy or new severe illness. 3. Intolerable toxicity. 4. Subject/investigator decision. 5. Other reasons hindering continued participation. 5. Investigational Drugs and Treatment Protocol
  1. Source of Investigational Drugs: Lactobacillus johnsonii and matching placebo* are provided by Hangzhou Yuanda Biopharmaceutical Co., Ltd.
  2. Treatment Regimens Subjects will receive the following designed anticancer therapies every 3 weeks (unless disease progression or unacceptable toxicity occurs). Concurrently, subjects will take oral Lactobacillus johnsonii (1*1011 CFU CFU, twice daily, dissolved in warm water) starting from the first anticancer treatment.

     Tumor-Specific Chemoimmunotherapy Protocols:

     Subgroup A: EGFR/ALK Wild-Type NSCLC (Unresectable/Metastatic)
* tislelizumab (200 mg IV on Day 1)
* pemetrexed (500 mg/m² BSA IV on Day 1)
* cisplatin (75 mg/m² BSA IV on Day 1). Subgroup B: PD-L1+ (CPS ≥1) Triple-Negative Breast Cancer (TNBC)
* Toripalimab (240 mg IV, Day 1)
* nab-paclitaxel (260 mg/m² BSA IV on Day 1)
* carboplatin (300 mg/m² BSA IV on Day 1) Subgroup C: HER2- Gastric/Gastroesophageal Junction Adenocarcinoma
* Tislelizumab (200 mg IV, Day 1)
* oxaliplatin (130 mg/m² BSA IV on Day 1)
* capecitabine (1000 mg/m² BSA orally twice daily, taken 30 minutes after meals on Days 1-14) 3. Investigational Drug Management Accountability: Drugs are strictly for trial use; no unauthorized redistribution. Designated staff must oversee storage, dispensing, returns, and destruction.

Documentation: Logistics records (shipment, receipt, allocation). Dispensing logs (recipient, verifier, date, dose, quantity). Reconciliation of unused drugs against prescriptions/records post-use.

Disposal: Unused drugs and packaging must be returned to the sponsor for destruction.

4. Permitted/Prohibited Concomitant Medications Allowed: Medications for non-excluded conditions (if stable at baseline). Prohibited: Antibiotics, other probiotics, herbal medicines, or CoQ10 (may interfere with Lactobacillus johnsonii assessment).

6. Study Procedures and Follow-up Plan Study Population: Patients with various tumors (lung cancer, breast cancer, gastric cancer) scheduled to receive immune checkpoint inhibitors. A total of 156 subjects will be enrolled across 4 medical centers (48 lung cancer, 52 breast cancer, 56 gastric cancer).

Screening Phase: Collection of medical history, demographic data, tumor stage/grade, pathological type, vital signs, physical examination, and pre-enrollment lab tests. Eligible subjects proceed to the treatment phase.

Treatment Phase: Daily administration of the study treatment per protocol. Scheduled visits for efficacy and safety assessments, including medication records, adverse events (AEs), and concomitant medications.

Follow-up Schedule:

* Timepoints: Baseline (Week 0), Weeks 6, 12, 18, and 24.
* Treatment regimen: Chemotherapy combined with immunotherapy (21-day cycles).
* Tumor response assessed every 2 cycles (42 days/6 weeks).
* Chemotherapy discontinued after 8 cycles (6 months).

Follow-up Assessments:

Biological samples: Fecal and plasma collection at Weeks 0, 6, 12, 18, and 24 for:

* Gut microbiota composition (e.g., Lactobacillus johnsonii colonization).
* Indole derivative concentrations.

Clinical evaluations:

* Tumor progression (RECIST criteria).
* Treatment-related adverse events (TRAEs).
* Concomitant medications.
* Quality of life (QoL) scores. 7. Study Endpoints

Primary Endpoint:

Progression-free survival (PFS): Time from randomization to tumor progression or death (whichever occurs first).

Secondary Endpoints:

1. Changes in gut microbiome composition in stool samples: qPCR and 16sRNA analysis of microbial composition, including Lactobacillus johnsonii, immunotherapy-related bacterial abundance, and microbial diversity.
2. Changes in immune cell subsets in blood, just like Tregs, MDSCs, CD8+ T cells.
3. Changes in blood levels of IL-6, IL-8, and other cytokines/chemokines.
4. Changes in blood indole derivatives, for example, indolepropionic acid.
5. Characterization of the tumor microenvironment in archived tumor samples.
6. Objective Response Rate (ORR): Proportion of patients with tumor shrinkage meeting predefined criteria and sustained for a minimum duration (CR + PR).
7. Disease Control Rate (DCR): Percentage of evaluable cases achieving response (PR+CR) or stable disease (SD).
8. Duration of Response (DOR): Time from first objective response to disease progression (PD) or death before PD, reflecting the durability of ORR.
9. Disease Control Rate (DCR): Percentage of evaluable cases achieving response (PR+CR) or stable disease (SD).
10. Overall Survival (OS): Time from randomization to death from any cause.
11. Percentage of patients with immune checkpoint inhibitor-related adverse events (irAEs).

8. Adverse Events (AEs) and Safety Monitoring

Definitions:

* Adverse Event (AE):Any untoward medical occurrence post-treatment, regardless of causality.
* Serious AE (SAE): Results in death, hospitalization, disability, or birth defects.
* Drug-related AE: At least a plausible causal relationship with the study drug.

AE Documentation:

1. Required fields in CRF:

   * AE name, onset date, severity (CTCAE grade).
   * Action taken (e.g., treatment interruption).
   * Causality assessment (related/unrelated).
   * Outcome (resolved, ongoing, fatal).
2. Reporting Standards:

   * Completeness: Include drug dosing, concomitant medications, and corrective measures.
   * Clarity: Avoid medical abbreviations.

Safety Measures:

* Site-specific emergency protocols (e.g., glucocorticoids for irAEs).
* Real-time AE reporting to the Data Safety Monitoring Board (DSMB). (9) Management of Serious Adverse Events (SAEs)

Immediate Actions:

Investigators must promptly implement appropriate and proactive rescue/protective measures for subjects experiencing SAEs and may decide to discontinue the study based on clinical judgment.

Reporting Requirements: All SAEs must be immediately reported in writing to the sponsor, followed by detailed written follow-up reports. Reports must use the subject's unique trial identification code (not personal identifiers such as name, ID number, or address).

Fatal Events: Additional documents (e.g., autopsy/final medical reports) must be submitted to the sponsor and ethics committee (EC).

Safety Information Handling: Investigators must promptly review safety updates from the sponsor, assess potential impacts on subject treatment, and communicate adjustments to subjects as needed. Suspected unexpected serious adverse reactions (SUSARs) must be reported to the EC and trial institution per sponsor-provided information.

Regulatory Compliance: Follow the *NMPA Standards and Procedures for Expedited Safety Reporting During Drug Clinical Trials. The sponsor must report all SUSARs (definitely or possibly drug-related) and other specified events to the National Medical Products Administration (NMPA) within mandated timelines.

(10) Data Management

Roles & Procedures:

* A professional data management team ensures accuracy, completeness, confidentiality, and traceability of trial data.
* Case Report Forms (CRFs):
* Completed by authorized personnel using source documents.
* Monitors verify CRF data against source records.
* Data Quality Control:
* Data managers check logic, authenticity, timeliness, and completeness.
* Queries are issued for discrepancies; investigators must respond promptly.

Database Locking:

* The database is locked after final approval by the sponsor, statistician, and data managers.
* Post-lock modifications require team consensus and must be fully documented. (11) Statistical Analysis

Analysis Plan (SAP):

* Drafted by statisticians after finalizing the protocol/CRFs; updated during the trial.
* Version-controlled and signed before database lock. Protocol amendments trigger SAP revisions.

Analysis Datasets:

1. Full Analysis Set (FAS): All randomized subjects receiving the study drug (primary efficacy analysis).
2. Per Protocol Set (PPS): Subjects compliant with the protocol.
3. Safety Set (SS): All subjects receiving ≥1 dose of the study drug.

Methods:

* Software: SPSS 26.0; significance threshold p<0.05 (two-tailed).
* Data Types:
* Continuous: Shapiro-Wilk test for normality → mean±SD (t-test) or median [IQR] (Mann-Whitney U).
* Categorical: Frequency (%) → Chi-square/Fisher's exact test.
* Longitudinal Data: Repeated-measures ANOVA or generalized estimating equations (GEE).
* Microbiome/Metabolites:
* α/β-diversity; differential abundance (Wilcoxon/t-test).
* Pearson correlation for clinical-microbiome/metabolite associations.
* Adverse Events:
* Coded via MedDRA; incidence rates compared using Fisher's exact test. (12) Study Management

To ensure subject rights protection, data accuracy, and protocol/regulatory compliance, the following measures will be implemented:

1. Monitoring

   * Qualified monitors will conduct **regular, systematic site visits to verify:
   * Protocol adherence
   * Consistency between reported data and source documents
   * Monitoring reports will document findings and escalate issues to the sponsor and investigators.
2. Audits & Inspections

   * Audits: Conducted by independent personnel (not directly involved in the trial).
   * Inspections: Initiated by regulatory authorities (e.g., NMPA).
   * Site obligations:
   * Provide direct access to source data/documents.
   * Notify the sponsor immediately upon regulatory inspection requests.
3. Training & Compliance - Investigator meetings must be held before trial initiation to:

   - Review the protocol, CRFs, and drug dispensing procedures.
   * Ensure uniform data collection/adjudication standards.
   * All site personnel must:
   * Complete GCP and protocol-specific training (records maintained).
   * Follow SOPs and GCP guidelines strictly.
4. Quality Control (QC) & Quality Assurance (QA)

   * Personnel qualifications:
   * Only GCP-trained physicians/researchers may participate.
   * Laboratory QC:
   * SOPs for lab assays + certified quality control (e.g., CAP/CLIA).
   * Monitoring:
   * CRF vs. source data verification.
   * Drug storage/accounting checks.
   * Confirmation of informed consent (IC) for all subjects.
   * Audits:
   * Conducted by independent, GCP-certified auditors to assess:
   * Protocol/SOP compliance.
   * Data integrity (timely, accurate, complete). （13）Ethical Requirements

<!-- -->

1. Regulatory Compliance

   * Follow NMPA GCP, Helsinki Declaration, and Chinese laws.
   * Protocol/amendments and IC forms require EC approval before implementation.
2. Investigator Eligibility

   * Exclude personnel with:
   * Disciplinary actions (e.g., revoked medical license).
   * History of academic fraud.
3. Informed Consent (IC) Process - Pre-study requirements:

   - Explain purpose, procedures, risks/benefits, and voluntary participation.

   - Emphasize:

   - Right to withdraw without penalty.

   - Alternative treatments available.

   - Confidentiality of records (accessible only to authorized parties).

   - Documentation:

   - Subjects must sign EC-approved IC forms before any study procedures.
   * Provide copies of signed IC forms to subjects.
4. Low-Risk Procedures

   * Minimally invasive tests (e.g., blood draws are classified as routine/low-risk.

If a subject (or legal representative) cannot read/write, the following steps must be followed:

- Impartial Witness Requirement: A neutral, independent witness (uninvolved in the trial) must participate in the entire IC process. The witness must observe the researcher's verbal explanation of the study (including risks, benefits, and rights)，confirm that all written information (IC form) was accurately read aloud and understood.

Documentation: After the subject (or representative) provides oral consent, the witness must: Sign and date the IC form (attesting to the subject's comprehension and voluntary participation). Note: The subject's thumbprint (or equivalent mark) may replace a signature if culturally appropriate. The researcher must also sign, confirming adherence to the process.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age 18-75 years.
3. Histologically confirmed unresectable/metastatic tumors:

   EGFR/ALK wild-type adenocarcinoma non-small cell lung cancer (NSCLC) PD-L1+ (CPS≥1) triple-negative breast cancer (TNBC) HER2- gastric/gastroesophageal adenocarcinoma
4. ≥1 measurable lesion (RECIST v1.1).
5. Progression after PD-1/PD-L1 inhibitor therapy (defined as:

   * ≥2 doses administred.
   * Radiographic progression per RECIST/iRECIST/irRECIST, confirmed ≥4 weeks later.
   * Progression within 12 weeks of last PD-1/PD-L1 dose.
6. Adequate organ function.
7. ECOG performance status 0-1.
8. Negative pregnancy test (urine/serum β-HCG) for women of childbearing potential.

Exclusion Criteria:

* 1. Prior allogeneic transplantation (cells, tissues, or solid organs). 2. History of immune-related adverse events (irAEs) from immunomodulators (e.g., PD-1/PD-L1 or CTLA-4 inhibitors) leading to permanent discontinuation or Grade 3/4 severity.

  3. Recent anticancer therapy (chemotherapy/immunotherapy/biologics/experimental drugs) within: <5 half-lives of the drug or <21 days before starting study treatment (whichever is shorter). Exceptions: Stable hormone therapy (e.g., for prostate/breast/ovarian cancer).

  4. Concomitant corticosteroid use (>10 mg prednisone/day or equivalent) within 7 days prior to treatment, unless for physiological replacement (≤10 mg/day) or non-immunosuppressive purposes (e.g., inhaled/topical steroids).

  5. Severe cardiac dysfunction, including: NYHA Class III-IV heart failure, symptomatic coronary artery disease, severe ventricular arrhythmias, myocardial infarction/unstable angina within 6 months.

  6. Active autoimmune disease requiring systemic treatment (immunosuppressants/corticosteroids) in the past 2 years, except: Hormone replacement (thyroxine, insulin, physiologic corticosteroids).

  7. Active severe infection requiring systemic therapy. 8. Antibiotic use completed within 2 weeks before the first dose. 9. Psychiatric or substance abuse disorders compromising protocol compliance. 10. Live vaccines administered within 28 days before treatment. 11. Active HIV or hepatitis (A/B/C) infection. 12. History of steroid-requiring (non-infectious) pneumonitis or current active pneumonitis.

  13. Other malignancies requiring active treatment or progressing within 2 years (exceptions: Non-melanoma skin cancer, cervical/prostate carcinoma in situ).

  14. Pregnancy or lactation. 15. Known intolerance/allergy to study drugs. 16. Other conditions deemed unsuitable by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the end of treatment at 24weeks
  Progression-Free Survival (PFS): Time from randomization to tumor progression or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints | From enrollment to the end of treatment at 24 weeks
  1. Changes in gut microbiome composition in stool samples: qPCR and 16sRNA analysis of microbial composition, including Lactobacillus johnsonii, immunotherapy-related bacterial abundance, and microbial diversity. 2. Changes in immune cell subsets in blood, just like Tregs, MDSCs, CD8+ T cells. 3. Changes in blood levels of IL-6, IL-8, and other cytokines/chemokines. 4. Changes in blood indole derivatives, for example, indolepropionic acid. 5. Characterization of the tumor microenvironment in archived tumor samples. 6. Objective Response Rate (ORR): Proportion of patients with tumor shrinkage meeting predefined criteria and sustained for a minimum duration (CR + PR). 7. Disease Control Rate (DCR): Percentage of evaluable cases achieving response (PR+CR) or stable disease (SD). 8. Duration of Response (DOR): Time from first objective response to disease progression (PD) or death before PD, reflecting the durability of ORR. 9. Disease Control Rate (DCR)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia DJ, Wang QW, Hu YY, He JM, Ge QW, Qi YD, Chen LY, Zhang Y, Fan LN, Lin YF, Sun Y, Jiang Y, Wang L, Fang YF, He HQ, Pi XE, Liu W, Chen SJ, Wang LJ. Lactobacillus johnsonii alleviates colitis by TLR1/2-STAT3 mediated CD206+ macrophagesIL-10 activation. Gut Microbes. 2022 Jan-Dec;14(1):2145843. doi: 10.1080/19490976.2022.2145843. PMID 36398889